CLINICAL TRIAL: NCT04397588
Title: Extracorporeal Membrane Oxygenation (ECMO) as a Therapeutic Option in Severe Form of COVID-19: a Nationwide Cohort Study
Brief Title: Extracorporeal Membrane Oxygenation (ECMO) and Coronavirus Disease (COVID) 19
Acronym: ECMO-SARS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC20_8979 ECMO-SARS
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-05

CONDITIONS: ARDS Related to Severe Acute Respiratory Syndrome-Coronavirus (SARS-CoV) 2; Acute Refractory Heart Failure Related to SARS-CoV 2
Keywords: ECMO; COVID-19; SARS-CoV2; ARDS; Myocarditis; Heart failure
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Myocarditis; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The role of ECMO in the treatment of patients with severe COVID-19 (Acute Respiratory Distress Syndrome (ARDS) and/or acute refractory heart failure) is not yet known. The present study will aim to report the results of the ECMO management of the most severe forms of COVID-19 through the first French ECMO registry.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the hospital survival of COVID-19 patients supported by venovenous or venoarterial ECMO in a multicenter registry.

The secondary objectives are to describe the characteristics of COVID-19 patients who have received ECMO support, to identify the risk factors associated with hospital mortality, to analyze the outcomes after ECMO weaning including survival at day 28 and day 90, and to analyze the utility of a circulatory support mobile unit in a severe pandemic

Inclusions are both prospective and retrospective in order to collect data over the whole pandemic

ELIGIBILITY:
Inclusion Criteria:

* All COVID-19 patients, adults or children,
* Tested positive by RT-PCR for SARS-CoV2 (nasopharyngeal swabs, sputum, endotracheal aspiration, bronchoalveolar lavage or stool sample) and / or with a diagnosis made on chest CT findings,
* Supported by venovenous or venoarterial ECMO

Exclusion Criteria:

* Temporary legally protected Adults over a set period or waiting for protection supervision, guardianship
* Patients or proxies who express their opposition to study participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill COVID-19 patients with ARDS or/and acute refractory heart failure
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2020-10-21 (Estimated); Study Completion 2020-10-21 (Estimated)

PRIMARY OUTCOMES:
Hospital mortality | up to 90 days
  Hospital mortality

SECONDARY OUTCOMES:
Mortality Day 28 | Day 28
  Mortality Day 28
Mortality Day 90 | Day 90
  Mortality Day 90
Ventilator-free days | Day 28
  Ventilator-free days
Intensive care unit-free days | Day 28
  ICU-free days
Hospital-free days | Day 28
  Hospital-free days

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Nesseler, doctor, Principal Investigator — Rennes University Hospital; André Vincentelli, professor, Principal Investigator — Lille University Hospital
Locations (44):
- France (44):
  - Angers University Hospital, Angers
  - Besançon Hospital, Besançon
  - Brest university Hospital, Brest
  - Caen University Hospital, Caen
  - Clermont ferrand University hospital, Clermont-Ferrand
  - APHP Henri Mondor Paris University Hospital, Créteil
  - Dijon University Hospital, Dijon
  - Vendée Hospital, La Roche-sur-Yon
  - Grenoble University Hospital, La Tronche
  - APHP Kremli Bicetre Paris University Hospital, Le Kremlin-Bicêtre
  - Marie Lannelongue Hospital, Le Plessis-Robinson
  - Lens Hospital, Lens
  - Lille University Hospital, Lille
  - Limoges University Hospital, Limoges
  - Clinique de la Sauvegarde, Lyon
  - Lyon University Hospital, Lyon
  - Marseille Européen Hospital, Marseille
  - APHM la Timone- Marseille University Hospital, Marseille
  - Clairval Hospital, Marseille
  - Metz University Hospital, Metz
  - Montpellier University Hospital, Montpellier
  - Emile Muller Hospital, Mulhouse
  - Nancy University Hospital, Nancy
  - Nantes University Hospital, Nantes
  - Ambroise Paré Hospital, Neuilly-sur-Seine
  - Nimes University Hospital, Nîmes
  - Institut Mutualiste Montsouris, Paris
  - APHP Hopital Européen Georges Pompidou - Paris University Hospital, Paris
  - APHP necker Paris University Hospital, Paris
  - APHP Bichat - Paris University Hospital, Paris
  - APHP La Pitié Salpêtrière Paris University Hospital, Paris
  - Bordeaux University Hospital, Pessac
  - Poitiers University hospital, Poitiers
  - Reims University hospital, Reims
  - Rennes University hospital, Rennes
  - Rouen University Hospital, Rouen
  - Saint brieuc Hospital, Saint-Brieuc
  - La Réunion University Hospital, Saint-Denis
  - Saint Etienne University Hospital, Saint-Etienne
  - Saint Nazaire Hospital, Saint-Nazaire
  - Strasbourg University Hospital, Strasbourg
  - Toulouse University Hospital - Rangueil Hospital, Toulouse
  - Tours University Hospital, Tours
  - Bretagne Atlantique Hospital, Vannes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nesseler N, Mansour A, Schmidt M, Para M, Porto A, Falcoz PE, Mongardon N, Fougerou C, Ross JT, Beurton A, Gaide-Chevronnay L, Guinot PG, Lebreton G, Flecher E, Vincentelli A, Massart N; ECMOSARS Investigators; SFAR Research Network. Healthcare-associated infections in patients with severe COVID-19 supported with extracorporeal membrane oxygenation: a nationwide cohort study. Crit Care. 2024 Feb 20;28(1):54. doi: 10.1186/s13054-024-04832-3. PMID 38374103
- [Derived] Massart N, Guervilly C, Mansour A, Porto A, Flecher E, Esvan M, Fougerou C, Fillatre P, Duburcq T, Lebreton G, Para M, Stephan F, Hraiech S, Ross JT, Schmidt M, Vincentelli A, Nesseler N; Extracorporeal Membrane Oxygenation for Respiratory Failure and/or Heart failure related to Severe Acute Respiratory Syndrome Coronavirus 2 (ECMOSARS) Investigators. Impact of Prone Position in COVID-19 Patients on Extracorporeal Membrane Oxygenation. Crit Care Med. 2023 Jan 1;51(1):36-46. doi: 10.1097/CCM.0000000000005714. Epub 2022 Nov 11. PMID 36519982
- [Derived] Mansour A, Flecher E, Schmidt M, Rozec B, Gouin-Thibault I, Esvan M, Fougerou C, Levy B, Porto A, Ross JT, Para M, Manganiello S, Lebreton G, Vincentelli A, Nesseler N; ECMOSARS Investigators. Bleeding and thrombotic events in patients with severe COVID-19 supported with extracorporeal membrane oxygenation: a nationwide cohort study. Intensive Care Med. 2022 Aug;48(8):1039-1052. doi: 10.1007/s00134-022-06794-y. Epub 2022 Jul 13. PMID 35829723